CLINICAL TRIAL: NCT06715488
Title: Automated Detection Methods for Inflammatory Arthritis and Formation of an Image Database
Brief Title: Automated Arthritis Detection Using Artificial Intelligence on Smartphone Photographs
Acronym: AISynovitis
Status: Active, not recruiting | Type: Observational
Sponsor: Med2Measure (Industry)
Collaborators: IISER Pune (Unknown)
Responsible Party: Sponsor
Other Study IDs: M2M-ID0001
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Rheumatoid Arthritis &Amp; Other Inflammatory Polyarthropathies; Peripheral Spondyloarthritis; Inflammatory Arthritis
Keywords: Artificial intelligence for arthritis diagnosis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inflammatory arthritis: Patients with inflammatory arthritis regardless of etiology including rheumatoid arthritis, psoriatic arthritis, systemic lupus erythematosis and viral arthritis
  Interventions: Diagnostic Test: AI assisted smartphone diagnosis

INTERVENTIONS:
Diagnostic Test: AI assisted smartphone diagnosis — Patients will examination and clinical photographs for convolutional networks to diagnose inflammatory arthritis

SUMMARY:
The investigators are testing the ability of convolutional neural networks (CNNs), that is artificial intelligence, on smartphone photographs in detecting inflammatory arthritis. This promises to be an efficient, accurate, and non-invasive diagnostic tool that will significantly improve early detection and management of inflammatory arthritis.

DETAILED DESCRIPTION:
Over the past 4 years the investigators have aimed to help the early detection of arthritis leveraging artificial intelligence. This project aims to detect arthritis based on smart phone photographs of joint areas that make it scalable and available in the community. This group first developed a compelling proof-of-concept pipeline and models using 100 patients. (published in Frontiers in Medicine, Nov 2023, wherein they demonstrated that this technology works with reasonable accuracy in the lab, viz Technology Readiness Level currently stands at 3-4). They followed with a newer paper (submitted for publication, available on preprint server MedRxiv) that trained two different CNNs, a screening CNN on uncropped hands that distinguishes patients from controls followed by joint specific detections.

The system involves supporting infrastructure that will enable efficient detection of arthritis. This includes

1. Collection of photos in a standardized manner using custom designed boxes
2. Using and testing a browser pipeline
3. The CNN models will be trained on the dataset of photographs taken in this and results will be deployed to doctors in the community. This ensures a doctor in the loop that can later take action on the results for further confirmatory tests or management.
4. Understanding knowledge, attitude of patients and doctors towards AI in clinical decision making algorithms

This is a Prospective, non-interventional study and this project only involves an investigator taking a smartphone photograph of some joint areas kept in standardized positions. This involves no risk to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Inflammatory arthritis of any etiology

Exclusion Criteria:

* Severe deformity that hampers standardization of photographs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with inflammatory arthritis. This can include but is not limited to rheumatoid arthritis, lupus, psoriatic arthritis, peripheral spondyloarthritis, viral arthritis.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of AI diagnosis against specialist (rheumatologist) opinion | 3 years
  Concordance of detection of synovitis by convolutional neural network (binary) with a clinically diagnosed specialist opinion (rheumatologist opinion)

SECONDARY OUTCOMES:
Accuracy of AI diagnosis against imaging diagnosis on Ultrasound | 3 years
  Concordance of detection of synovitis by convolutional neural network (binary) compared to musculoskeletal ultrasound
Sensitivity to change | 3 years
  Can the convolutional neural network detect change from an inflamed to an non-inflamed joint

CONTACTS AND LOCATIONS:
Overall Officials: Sanat Phatak, MD, DM, Principal Investigator — Med2Measure
Locations (2):
- India (2):
  - Rheumatology Clinic, Pune, Maharashtra
  - Poona Superspeciality Clinic, Pune

IPD SHARING:
Plan to Share IPD: Yes
Deidentified photographs and clinical information excluding HIPAA variables
Supporting Information: Study Protocol, ICF, CSR
Time Frame: January 2027-January 2028
Access Criteria: Researchers with a scientific plan can get in touch with the principal investigator with a brief note.